CLINICAL TRIAL: NCT02648074
Title: Eosinophil Induced Airway Smooth Muscle Remodelling in Asthma
Brief Title: Eosinophil Induced Remodelling in Asthma
Acronym: ERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Research Council of Lithuania (Other); University of Groningen (Other)
Responsible Party: Principal Investigator, Kestutis Malakauskas, Prof. dr., Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MIP-010/2014; PSUL-010/2014 (Other: Lithuanian University of Health Sciences)
Record Dates: First submitted 2015-12-21; First posted 2016-01-06 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Allergic Asthma; Airway Remodelling
Keywords: asthma; eosinophils; airway smooth muscle; airway remodelling; integrins; cytokines
MeSH Terms: conditions — Airway Remodeling; Asthma | interventions — Allergens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergic asthma (Experimental): Bronchial asthma and sensitization to D. pteronyssinus allergen Interventions: Bronchial challenge with allergen; Eosinophil and linear bronchial smooth muscle cell co-culture formation.
  Interventions: Procedure: Bronchial challenge with allergen; Other: Co-culture formation
- Healthy subjects (Active Comparator): Healthy subjects without allergic and other chronic respiratory diseases (control group).
  Interventions: Bronchial challenge with allergen; Eosinophil and linear bronchial smooth muscle cell co-culture formation.
  Interventions: Procedure: Bronchial challenge with allergen; Other: Co-culture formation

INTERVENTIONS:
Procedure: Bronchial challenge with allergen — Bronchial challenge is performed with D. pteronyssinus allergen.
Other: Co-culture formation — Eosinophil and linear bronchial smooth muscle cell co-culture formation. Airway smooth muscle cell proliferation, eosinophil adhesion to the bronchial smooth muscle cells, the role of eosinophil integrins in the airway remodelling process is assessed in individual formed co-culture

SUMMARY:
Asthma is a chronic, inflammatory disease of the lung characterized by intermittent airway obstruction, airway hyperresponsiveness, presence of activated inflammatory cells, inflammatory mediators, and airway structural changes. Airway smooth muscle (ASM) cells actively participate in the remodelling and inflammatory processes through proliferation, release of proinflammatory cytokines, chemokines, and extracellular matrix (ECM) proteins. Eosinophils as essential inflammatory cells may be of importance in ASM remodelling. It is known that eosinophil induces ASM cells proliferation via the secretion of cysteinyl leukotrienes in asthmatics. However there is a possible direct eosinophil-ASM cells functional interaction by adhesion processes. It has been shown that integrins modulate ASM proliferation and contractile protein expression demonstrating allergen-induced ASM remodelling in an animal model of allergic asthma.

Wingless/integrase-1 (WNT) signaling regulates not only a wide range of developmental processes, but its aberrant activation can lead to disease. Recently, it was confirmed that genes polymorphisms in the WNT signaling pathway are associated with impaired lung function in childhood asthma. It was also found for the first time a relevant role of noncanonical WNT signaling in TGFβ-induced ECM expression by ASM cells and identified WNT-5A is the most abundant WNT ligand with increased expression in asthmatics. It demonstrates that WNT-5A could contribute to remodelling of the airways. Unfortunately, the effect of eosinophil on WNT secretion by ASM cells at present is unknown.

Despite the widely acknowledged significance of eosinophils in asthma pathogenesis, the mechanism of eosinophil induced ASM remodelling is unsolved.

DETAILED DESCRIPTION:
Asthma is a chronic, inflammatory disease of the lung characterized by intermittent airway obstruction, airway hyperresponsiveness, presence of activated inflammatory cells, inflammatory mediators, and remodeling in the airway. Airway remodeling characterizes as the cellular and structural changes in the airways, mainly resulting from repair processes in response to persistent inflammation. It is generally accepted that airway remodeling is closely related to the progression of airway hyperresponsiveness and the severity of asthma. The structural changes in the airway include airway smooth muscle (ASM) hypertrophy and hyperplasia, collagen deposition to the sub-epithelial basement membrane, hyperplasia of goblet cells, thickening of the airway mucosa and an increase in vascularity (Aceves and Broide, 2008).

Airway remodelling mostly is derived from airway inflammation, where eosinophils play a key role. The effect of intact eosinophils on ASM cells within a physiological context first time was investigated by Halwani with colleagues (2013). They found that prevention contact of eosinophils with ASM cells using specific antibodies or blocking cysteinyl leukotrienes was associated with inhibition of ASM proliferation in asthmatics. Moreover, Fanat et al. (2009) demonstrated that ASM-derived cytokines directly affect the eosinophils differentiation and maturation from progenitor cells, which can maintain airway eosinophilic inflammation and consequently the tissue remodelling in asthma. Furthermore, eosinophil deficient mice are protected from airway remodeling including collagen deposition and smooth muscle thickening (Humbles et al Science 2004, 305:1776-9).

Eosinophils seem to contribute to airway remodelling in several ways, including through release of eosinophil-derived mediators such as transforming growth factor (TGF)-β, secretion of cationic proteins, and cytokines, as well as through interactions with inflammatory and structural cells (Kariyawasam and Robinson, 2007; Aceves and Broide, 2008; Venge, 2010). Eosinophil-derived cytokines are in the modulation of Th2 responses that trigger macrophage production of TGF-β1, which serves as a stimulus for extracellular matrix (ECM) production (Fanta et al., 1999; Holgate, 2001). Masu et al. (2002) confirmed the proliferative effects of eosinophils lysates isolated from healthy donors on ASM cells. However, there is a possible direct eosinophil-ASM cells functional interaction by adhesion processes. Interaction of cells is mediated through integrins, a group of heterodimeric transmembrane glycoproteins (Hynes, 2002). Each integrin interacts or potentially interacts with counter-receptors on other cells or ligands deposited as part of the ECM (Humphries et al., 2006). The communication between eosinophil and ASM cells is not fully understood. Several integrins are expressed by eosinophils (α4β1, α6β1, αLβ2, αMβ2, αXβ2, αDβ2, α4β7) and ASM cell (α1β1, α2β1, α3β1, α4β1, α5β1, α6β1, α6β4, α7β1, α8β1, α9β1, αvβ1, αvβ3, αvβ5) (Teoh at al., 2012; Johansson and Mosher, 2013). It has been shown that integrins modulate ASM proliferation and contractile protein expression demonstrating allergen-induced ASM remodeling in an animal model of allergic asthma (Bart et al., 2010). Furthermore, several ASM derived integrins can function to activate latent TGF-beta into active TGF-beta in asthmatic airway smooth muscle (Tatler et al J Immunol 2011, 187:6094-107). Eosinophil integrins have the potential to mediate adhesion to endothelium in asthma (Barthel et al., 2008). Further studies indicate that integrins mediate trafficking of eosinophils to the lung and persistence in the ECM of the bronchi in models of allergen-induced acute and chronic asthma (Banerjee et al., 2007, 2009).

Wingless/integrase-1 (WNT) signalling regulates not only a wide range of developmental processes, but its aberrant activation can lead to disease. Up-regulation of several members of the WNT signalling pathway in the lungs of patients with idiopathic pulmonary fibrosis and other interstitial lung diseases has been demonstrated (Selman et al., 2006; Königshoff et al., 2008). More recently, Sharma et al. (2010) have confirmed that genes polymorphisms in the WNT signalling pathway are associated with impaired lung function in childhood asthma. Kumawat et al. (2013) for the first time reported a relevant role of noncanonical WNT signalling in TGFβ-induced extracellular matrix (ECM) expression by ASM cells and identified WNT-5A is the most abundant WNT ligand in ASM cells with increased expression in asthmatics. This is in line with Choy et al. (2011) who report that airway biopsies from Th2 high asthma patients have increased WNT-5A expression. Higher expression of WNT-5A in ASM cells demonstrates that WNT-5A could contribute to remodelling of the airways. Despite the reported role of WNT in airway remodelling, the regulation of WNT secretion by eosinophils or by eosinophil-ASM interactions is at present unknown.

Despite the widely acknowledged significance of eosinophils in asthma pathogenesis, the mechanism for eosinophil mediated airway remodeling is unsolved. At present understanding of eosinophils interaction and effect on ASM cells in asthma remains elusive. Therefore the nature of the interplay between these two cells types and the consequence of it needs to be investigated.

The aim of the Project: to assess the eosinophil mediated airway remodeling in asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18-50 years;
2. Allergic asthma and sensitization to house dust mites (D. pteronyssinus) allergen, approved with:

   2.1. Medical history and symptoms more than one year and 2.2. skin prick test positive for D. pteronyssinus (positive wheals are those exceeding 3mm in diameter greater than the negative control) and 2.3. Positive bronchial challenge with methacholine or documented completely reversible bronchial obstruction;
3. Stable lung function (FEV1≥70 perc.);
4. Postmenopausal women. Premenopausal women if pregnancy test is negative and they agree to use an effective contraceptive measures during the study;
5. Healthy subjects without allergic and other chronic respiratory diseases (control group);
6. Non- smokers;
7. Participants who gave his/her informed written consent.

Exclusion Criteria:

1. Asthma exacerbation 1 month prior to study
2. Clinically significant permanent allergy symptoms (ex. cat or dog dander induced allergy)
3. Contraindications to perform an allergy skin test and/or bronchial provocation test 3.1. Active airway infection 1 month prior the study; 3.2. Used medicaments: 3.2.1. Inhaled glucocorticoids intake 1 month prior the study; 3.2.2. Antihistamines intake 7 days prior the study; 3.2.3. Short acting β2 agonists 12 hours prior the study; 3.2.4. Long acting β2 agonists 2 days prior the study; 3.2.5. Leukotriene receptor antagonists prior 14 days;
4. If the histamine mean wheal diameter is <= 3 mm or control mean wheal diameter is >= 3 mm;
5. Contraindications for epinephrine;
6. Other significant mental and / or internal diseases and conditions, which could be as exclusion criteria due to the opinion of the researcher;
7. Alcohol or narcotic abuse;
8. Pregnancy;
9. Breast-feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Eosinophils and bronchial smooth muscle cell adhesion change assessment | In 30, 45, 60, 120, 240 minutes time points after eosinophils and bronchial smooth muscle cell interactions start
  There are used the individual eosinophil and airway smooth muscle cell co-culture. It is compared the strength of eosinophil adhesion to the bronchial smooth muscle cells in patients with asthma and healthy.
Bronchial smooth muscle cell proliferation change assessment by cell viability | In 48 and 72 hrs time points after eosinophils and linear bronchial smooth muscle co-culture formation
  Bronchial smooth muscle cell proliferation is assessed by cell viability

SECONDARY OUTCOMES:
The change of capacity of eosinophils' integrins to inhibit the bronchial smooth muscle cell proliferation in patients with asthma | In 48 and 72 hrs time points after eosinophils and linear bronchial smooth muscle co-culture formation
  Using the same eosinophils and linear bronchial smooth muscle cell culture, but in this measure is added integrins
The change of eosinophils' integrins interaction with bronchial smooth muscle cells and Wnt-5A protein production after allergen challenge | Up to 72 hrs time points after eosinophils (collected from blood of patients before and after bronchial provocation with an allergen) and linear bronchial smooth muscle co-culture formation
  The results are compared with the before and after bronchial provocation with Dermatophagoides pteronyssinus allergen. It is measured the integrins as specific adhesion molecules attachments to the bronchial smooth muscle cells after allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Kestutis Malakauskas, Prof., dr., Study Chair — Lithuanian University of Health Sciences, Pulmonology and Immunology Department
Locations (1):
- Lithuanian University of Health Sciences, Pulmonology and Immunology Department, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Januskevicius A, Gosens R, Sakalauskas R, Vaitkiene S, Janulaityte I, Halayko AJ, Hoppenot D, Malakauskas K. Suppression of Eosinophil Integrins Prevents Remodeling of Airway Smooth Muscle in Asthma. Front Physiol. 2017 Jan 9;7:680. doi: 10.3389/fphys.2016.00680. eCollection 2016. PMID 28119625
- [Derived] Januskevicius A, Vaitkiene S, Gosens R, Janulaityte I, Hoppenot D, Sakalauskas R, Malakauskas K. Eosinophils enhance WNT-5a and TGF-beta1 genes expression in airway smooth muscle cells and promote their proliferation by increased extracellular matrix proteins production in asthma. BMC Pulm Med. 2016 Jun 13;16(1):94. doi: 10.1186/s12890-016-0254-9. PMID 27297409